CLINICAL TRIAL: NCT06391346
Title: Evaluation of Gluteal Muscle Perfusion in Patients With Intermittent Gluteal Claudication by Non-invasive Multispectral Optoacoustic Tomography With Pre-post Study Design
Brief Title: Investigation of the Perfusion of Gluteal Muscle in Patients With Intermittent Gluteal Claudication by Non-invasive MSOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ulrich Rother (Other)
Responsible Party: Sponsor-Investigator, Ulrich Rother, PD Dr. med., University Hospital Erlangen
Organization: University Hospital Erlangen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MSOT-gluteal
Record Dates: First submitted 2024-02-20; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Peripheral Vascular Diseases; Peripheral Arterial Disease; Intermittent Claudication; Gluteal Claudication
Keywords: Peripheral Vascular Diseases; Peripheral Arterial Disease; Peripheral Artery Disease; PAD; Gluteal claudication; Buttock claudication; MSOT; Multispectral Optoacoustic Tomography
MeSH Terms: conditions — Peripheral Vascular Diseases; Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Intervention Model Description: Perfusion parameters from MSOT would be measured on patients with gluteal claudication in Fontain stage 2 before and after the revascularisation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient (Experimental): Multispectral Optoacoustic Tomography (MSOT) and B-Mode Ultrasound of the Musculus gluteus of the affected leg in PAD patients in Fontaine stage II (intermittent claudication)
  Physical assessment: Pulse status / Color-Coded Duplex Sonography / Ankle-Brachial Index / treadmill test / stepper exercise 2 minutes
  Interventions: Diagnostic Test: MSOT

INTERVENTIONS:
Diagnostic Test: MSOT — Non-invasive transcutaneous imaging of muscle components via infrared and near-infrared laser pulses

SUMMARY:
The objective of the proposed study is to define independent parameters for the diagnostic assessment of the perfusion situation of the gluteal muscle based on multispectral optoacoustic tomography (MSOT) in patients with gluteal claudication in Fontaine stage II (intermittent claudication) pre and post-intervention.

DETAILED DESCRIPTION:
This is a monocentric, prospective study which aims to exanimate the optoacoustic signals in gluteal muscle after a exercise in patients with PAD in Fontaine stage II before and after the revascularisation to verify the change of MSOT by improved vascularization. MSOT data will be correlated with CCDS, ABI, treadmill test, subjectively perceived absolute walking distance in everyday life, PAD-related life quality (VASCUQOL-6) and TASC II classification in angiographic imaging (only in case angiographic imaging is available and independent from this study).

Patients with gluteal claudication in Fontaine stage II will be recruited during the consulting hours of the Department of Vascular Surgery, University Hospital Erlangen. Following detailed information about the study and after providing written consent, relevant clinical data will be collected from the electronical patient file, if available. In addition, a thorough anamnesis interview for relevant data and CCDS would be performed. Afterwards, the MSOT parameters will be recorded on gluteal muscles before and after a stepper exercise two minutes or until the occurrence of claudication pain in the gluteal muscle. The more affected side is examined. All data will be adequately pseudonymized in compliance with data protection regulations before they are used for statistical analysis. The duration of the study for participants will be max. 90 minutes. The angiographic imaging will be reviewed and analyzed.

ELIGIBILITY:
Inclusion Criteria:

• Patient with gluteal claudication in Fontaine stage II and corresponding stenosis (common iliac artery, internal iliac artery or distal aorta)

Exclusion Criteria:

* Patients with PAD in Fontaine stage I, III and IV or Rutherford category 0, 4, 5 and 6 or healthy volunteers with diabetes mellitus, chronic renal failure, claudication symptoms, abnormal ABI or non-palpable foot pulses
* People with age under 18
* Absence of written consent
* Safety concerns of the study physician (person with physical, mental or psychiatric conditions which, by the judgement of the study physician, would compromise the person's safety or the quality of the data, thereby rendering the person an ineligible candidate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-23 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Optimal diagnostic MSOT thresholds | twice (before and after the intervention, up to two weeks)
  optimal diagnostic threshold for hemoglobin-associated MSOT parameters in gluteal muscle tissue in patients with intermittent claudication before and after exercise
Improvement of the MSOT parameters after the revascularisation | twice (before and after the intervention, up to two weeks)
  Change of hemoglobin-associated MSOT parameters in gluteal muscle tissue in patients with intermittent claudication before and after exercise after the revascularisation

SECONDARY OUTCOMES:
Difference between the corresponding MSOT values before and after exercis | twice (before and after the intervention, up to two weeks)
  Difference of the values before and after exercise for hemoglobin-associated parameters derived by transcutaneous MSOT in patients with gluteal claudication
Reperfusion profiles for hemoglobin-associated parameters | twice (before and after the intervention, up to two weeks)
  Curves of hemoglobin-associated MSOT parameters in the first ten minutes after exercise
Correlation of acquired MSOT parameters with the CCDS flow profile and PSV | single time point
  Hemoglobin-associated MSOT parameters in patients with gluteal claudication correlated with the flow profile and PSV of A. femoralis communis and A. poplitea determined by CCDS
Correlation of acquired MSOT parameters with the ABI | twice (before and after the intervention, up to two weeks)
  Hemoglobin-associated parameters derived by transcutaneous MSOT correlated with the ABI
Correlation of acquired MSOT parameters with threadmill test | twice (before and after the intervention, up to two weeks)
  Hemoglobin-associated MSOT parameters (units: arbitrary units (a.u.)) derived by transcutaneous MSOT correlated with Threadmill test
Correlation of acquired MSOT parameters with subjectively perceived maximum walking distance in everyday life | twice (before and after the intervention)
  hemoglobin-associated MSOT parameters (units: arbitrary units (a.u.)) derived by transcutaneous MSOT correlated with the subjectively perceived maximum walking distance in everyday life
Correlation of acquired MSOT parameters with the perceived PAD-specific quality of life (VASCUQOL-6 questionnaire) | twice (before and after the intervention, up to two weeks)
  hemoglobin-associated MSOT parameters (units: arbitrary units (a.u.)) derived by transcutaneous MSOT correlated with the perceived PAD-specific quality of life (VASCUQOL-6 questionnaire)
Correlation of acquired MSOT parameters with the TASC-classification (angiography) | twice (before and after the intervention, up to two weeks)
  hemoglobin-associated MSOT parameters (units: arbitrary units (a.u.)) derived by transcutaneous MSOT in patients with PAD in Fontaine stage II correlated with the TASC-classification (angiography)
Confounder analysis | twice (before and after the intervention, up to two weeks)
  Correlation of all collected parameters (anamnestic, demographic, physiological) with regard to their characteristics as basic confounders for the MSOT technique

CONTACTS AND LOCATIONS:
Locations (1):
- University of Erlangen-Nuremberg (FAU), Department of Vascular Surgery, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lawall H, Diehm C, Hoffmann U, Reinecke H. [Update PAVK: Epidemiology, comorbidity and prognosis of peripheral arterial obstructive disease]. Dtsch Med Wochenschr. 2015 Dec;140(24):1798-802. doi: 10.1055/s-0041-107064. Epub 2015 Dec 1. German. PMID 26625226
- [Result] Alpert JS, Larsen OA, Lassen NA. Exercise and intermittent claudication. Blood flow in the calf muscle during walking studied by the xenon-133 clearance method. Circulation. 1969 Mar;39(3):353-9. doi: 10.1161/01.cir.39.3.353. No abstract available. PMID 4885945
- [Result] Karlas A, Masthoff M, Kallmayer M, Helfen A, Bariotakis M, Fasoula NA, Schafers M, Seidensticker M, Eckstein HH, Ntziachristos V, Wildgruber M. Multispectral optoacoustic tomography of peripheral arterial disease based on muscle hemoglobin gradients-a pilot clinical study. Ann Transl Med. 2021 Jan;9(1):36. doi: 10.21037/atm-20-3321. PMID 33553329
- [Result] Larsen ASF, Reiersen AT, Jacobsen MB, Klow NE, Nordanstig J, Morgan M, Wesche J. Validation of the Vascular quality of life questionnaire - 6 for clinical use in patients with lower limb peripheral arterial disease. Health Qual Life Outcomes. 2017 Sep 22;15(1):184. doi: 10.1186/s12955-017-0760-3. PMID 28938901
- [Result] Abraham P, Picquet J, Vielle B, Sigaudo-Roussel D, Paisant-Thouveny F, Enon B, Saumet JL. Transcutaneous oxygen pressure measurements on the buttocks during exercise to detect proximal arterial ischemia: comparison with arteriography. Circulation. 2003 Apr 15;107(14):1896-900. doi: 10.1161/01.CIR.0000060500.60646.E0. Epub 2003 Mar 31. PMID 12668524
- [Result] Assi H, Cao R, Castelino M, Cox B, Gilbert FJ, Grohl J, Gurusamy K, Hacker L, Ivory AM, Joseph J, Knieling F, Leahy MJ, Lilaj L, Manohar S, Meglinski I, Moran C, Murray A, Oraevsky AA, Pagel MD, Pramanik M, Raymond J, Singh MKA, Vogt WC, Wang L, Yang S, Members Of Ipasc, Bohndiek SE. A review of a strategic roadmapping exercise to advance clinical translation of photoacoustic imaging: From current barriers to future adoption. Photoacoustics. 2023 Aug 2;32:100539. doi: 10.1016/j.pacs.2023.100539. eCollection 2023 Aug. PMID 37600964
- [Result] Audonnet M, Signolet I, Colas-Ribas C, Ammi M, Abraham P, Henni S. Exercise Transcutaneous Oximetry of the Buttocks - External Validation With Computed Tomography Angiography. Circ J. 2017 Jul 25;81(8):1123-1128. doi: 10.1253/circj.CJ-16-1316. Epub 2017 Apr 13. PMID 28413177
- [Result] Batt M, Baque J, Bouillanne PJ, Hassen-Khodja R, Haudebourg P, Thevenin B. Percutaneous angioplasty of the superior gluteal artery for buttock claudication: a report of seven cases and literature review. J Vasc Surg. 2006 May;43(5):987-91. doi: 10.1016/j.jvs.2006.01.024. PMID 16678694
- [Result] Gernigon M, Marchand J, Ouedraogo N, Leftheriotis G, Piquet JM, Abraham P. Proximal ischemia is a frequent cause of exercise-induced pain in patients with a normal ankle to brachial index at rest. Pain Physician. 2013 Jan;16(1):57-64. PMID 23340534